CLINICAL TRIAL: NCT04071314
Title: Evaluating the Alimentary and Respiratory Tracts in Health and Disease (EARTH) Research Program.
Acronym: EARTH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Dr Michael Coffey, Principal Investigator, The University of New South Wales
Other Study IDs: HREC/18/SCHN/26
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cystic Fibrosis; Hirschprung's Disease; Obstructive Sleep Apnea; Healthy
Keywords: Microbiota; Gastrointestinal Microbiome; Diet; Signs and Symptoms; Quality of Life; Anxiety; Depression
MeSH Terms: conditions — Cystic Fibrosis; Sleep Apnea, Obstructive; Signs and Symptoms; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A stool sample;
  * An oropharyngeal swab or sputum sample (a sputum sample will be obtained in children able to expectorate and an oropharyngeal swab will be collected in children unable to expectorate).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cystic fibrosis: Children diagnosed with cystic fibrosis. Children aged between 0 and 18 years.
- Hirschsprung's disease: Children diagnosed with Hirschsprung's disease. Children aged between 0 and 18 years.
- Obstructive sleep apnoea: Children diagnosed with obstructive sleep apnoea. Children aged between 0 and 18 years.
- Healthy controls: Children free of any chronic health condition. Children aged between 0 and 18 years.

SUMMARY:
The investigators have established the "Evaluating the Alimentary and Respiratory Tracts in Health and disease" (EARTH) research program. It provides a structured approach to analysing gastrointestinal and respiratory microbiomes, along with diet and symptomatology, in children with a gastrointestinal and/or respiratory condition with recognised long-term morbidity (e.g. cystic fibrosis, obstructive sleep apnoea, or Hirschsprung's disease).

The EARTH program consists of a series of prospective, longitudinal, controlled, observational studies, with each individual study comparing children with a chronic gastrointestinal and/or respiratory condition to healthy controls (HC). It will be conducted in an Australian tertiary paediatric hospital (although the methodology is applicable to other settings). Children with a chronic gastrointestinal and/or respiratory condition will be compared to age and gender matched HC across a 12-month period. The following will be collected at baseline, 6 and 12 months: (i) a stool sample, (ii) an oropharyngeal swab or sputum sample, (iii) a semi-quantitative food frequency questionnaire, (iv) details of disease symptomatology, (v) health-related quality of life, and (vi) psychosocial factors. Data on the intestinal and respiratory microbiomes and diet will be compared between children with a condition and HC. Correlations between dietary intake (energy, macro- and micro-nutrients), intestinal and respiratory microbiomes within each group will be explored. Data on disease symptomatology, quality of life and psychosocial factors will also be compared between children with a condition and HC.

The investigators hypothesise that:

(i) Children with chronic gastrointestinal and/or respiratory conditions will have altered intestinal and respiratory microbiomes compared to healthy children, and (ii) Diet plays a key role in influencing the intestinal and respiratory microbiomes and this may impact on clinical outcomes, biomarkers of disease, and health-related quality of life.

DETAILED DESCRIPTION:
The objective of this research program is to evaluate and compare children with a chronic gastrointestinal and/or respiratory condition and age and gender matched HC. The primary objectives include analysing the intestinal and respiratory microbiomes (using an integrated "omics" approach) and dietary intake using validated, food frequency quetsionnaires. The secondary objectives include evaluating:

1. Known inflammatory biomarkers.
2. Symptomatology and health-related quality of life (HRQOL) using validated measures.
3. Phenotypic and clinical information.
4. Sociodemographic factors Additional secondary objectives include correlating within children with the same condition: (i) dietary intake with the intestinal microbiome; (ii) dietary intake with the respiratory microbiome; and (iii) the intestinal and respiratory microbiomes.

The investigators hypothesise that:

(i) Children with chronic gastrointestinal and/or respiratory conditions will have altered intestinal and respiratory microbiomes compared to healthy children, and (ii) Diet plays a key role in influencing the intestinal and respiratory microbiomes and this may impact on clinical outcomes, biomarkers of disease, and health-related quality of life.

To our knowledge, this program will enable the first series of studies comparing the intestinal and respiratory microbiomes and diet in children with chronic gastrointestinal and/or respiratory conditions. Initial results will be hypothesis-generating and used to direct future studies tailored to a specific focus or line of inquiry. Additionally, studies from this research program have potential for direct translation into clinical care as diet is a highly modifiable factor.

Study design. The EARTH program provides a framework for a series of prospective, longitudinal, controlled, observational studies, with each individual study comparing children with a chronic gastrointestinal and/or respiratory condition to HC. A single healthy control group will be used for comparison against all conditions. The standardised methodological approach will also allow for comparisons between different health conditions.

Procedures.

Each participant will be assessed on three occasions over a 12-month period; at study entry, 6- and 12-month follow-up. At each time-point, the following will be collected:

* A stool sample;
* An oropharyngeal swab or sputum sample (a sputum sample will be obtained in children able to expectorate and an oropharyngeal swab will be collected in children unable to expectorate);
* Dietary intake measured using the Australian Child and Adolescent Eating Survey (ACAES) (2 to 18 years) or 24-hour food recall (0 up to 2 years);
* A secure, password-protected online survey comprising:

  i. PedsQL Infant Scales (0-2yr) & Gastrointestinal Symptoms Module (2-18yr),41-43 tailored to age; ii. Rome IV Questionnaire (0 to 18 years); iii. Spence Children's Anxiety Scale (3 to 18 years); iv. Short Mood and Feelings Questionnaires (6 to 18 years); v. Clinical and biochemical results obtained through routine care and hospitalisations (if available); vi. Sociodemographic factors (baseline survey only);
* Anthropometrics: height, weight and BMI z-scores.

ELIGIBILITY:
Inclusion Criteria:

* Are aged between 0 and 18 years;
* Have been diagnosed with a chronic gastrointestinal and/or respiratory condition defined by consensus diagnostic criteria; or
* Are free of any chronic health condition (healthy control group); and
* Have a parent(s)/carer(s) who provides informed consent, or are at least 16 years old and provide informed consent.

Exclusion Criteria:

* Children who have an unrelated coexisting chronic medical illness(es) associated with alterations in dietary intake or suspected alterations in the intestinal and/or respiratory microbiomes;
* Inability to comply with study requirements;
* Parent(s)/guardian(s) are unable to speak English or do not have a reading level age of at least 12 years.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Studies will be carried out at a single centre; the Sydney Children's Hospital (SCH) in Randwick, Australia. SCH is a tertiary paediatric hospital. Participants with chronic gastrointestinal and/or respiratory conditions will be approached at their routine clinic appointments in the outpatient department. Flyers will be placed in the hospital for recruitment of HC.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2023-03-13 (Estimated); Study Completion 2023-03-13 (Estimated)

PRIMARY OUTCOMES:
1A.i.0 Intestinal Microbiome (Bacteria) - Richness | Baseline
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.i.6 Intestinal Microbiome (Bacteria) - Richness | Change from baseline at 6 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.i.12 Intestinal Microbiome (Bacteria) - Richness | Change from baseline at 12 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.ii.0 Intestinal Microbiome (Bacteria) - Shannon index | Baseline
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.ii.6 Intestinal Microbiome (Bacteria) - Shannon index | Change from baseline at 6 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.ii.12 Intestinal Microbiome (Bacteria) - Shannon index | Change from baseline at 12 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.iii.0 Intestinal Microbiome (Bacteria) - UNIFRAC distances | Baseline
  Measurement of beta diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.iii.6 Intestinal Microbiome (Bacteria) - UNIFRAC distances | 6 months
  Measurement of beta diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.iii.12 Intestinal Microbiome (Bacteria) - UNIFRAC distances | 12 months
  Measurement of beta diversity (assessed using 16S rRNA or metagenomic gene sequencing).
1A.iv.0 Intestinal Microbiome (Bacteria) - relative abundances of bacteria | Baseline
  ANCOM analysis (assessed using 16S rRNA or metagenomic gene sequencing).
1A.iv.6 Intestinal Microbiome (Bacteria) - relative abundances of bacteria | Change from baseline at 6 months
  ANCOM analysis (assessed using 16S rRNA or metagenomic gene sequencing).
1A.iv.12 Intestinal Microbiome (Bacteria) - relative abundances of bacteria | Change from baseline at 12 months
  ANCOM analysis (assessed using 16S rRNA or metagenomic gene sequencing).
1B.i.0 Intestinal Microbiome (Proteome) - normalised abundances of proteins | Baseline
  (assessed using LC-MS).
1B.i.6 Intestinal Microbiome (Proteome) - normalised abundances of proteins | Change from baseline at 6 months
  (assessed using LC-MS).
1B.i.12 Intestinal Microbiome (Proteome) - normalised abundances of proteins | Change from baseline at 12 months
  (assessed using LC-MS).
1C.i.0 Intestinal Microbiome (Metabolome) - normalised abundances of metabolites | Baseline
  (assessed using LC-MS).
1C.i.6 Intestinal Microbiome (Metabolome) - normalised abundances of metabolites | Change from baseline at 6 months
  (assessed using LC-MS).
1C.i.12 Intestinal Microbiome (Metabolome) - normalised abundances of metabolites | Change from baseline at 12 months
  (assessed using LC-MS).
1D.i.0 Intestinal Microbiome (Viruses) - Richness | Baseline
  Measurement of alpha diversity (assessed metagenomic sequencing).
1D.i.6 Intestinal Microbiome (Viruses) - Richness | Change from baseline at 6 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
1D.i.12 Intestinal Microbiome (Viruses) - Richness | Change from baseline at 12 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
1D.ii.0 Intestinal Microbiome (Viruses) - Shannon index | Baseline
  Measurement of alpha diversity (assessed metagenomic sequencing).
1D.ii.6 Intestinal Microbiome (Viruses) - Shannon index | Change from baseline at 6 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
1D.ii.12 Intestinal Microbiome (Viruses) - Shannon index | Change from baseline at 12 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
1D.iii.0 Intestinal Microbiome (Viruses) - Bray-Curtis dissimilarity | Baseline
  Measurement of beta diversity (assessed metagenomic sequencing).
1D.iii.6 Intestinal Microbiome (Viruses) - Bray-Curtis dissimilarity | 6 months
  Measurement of beta diversity (assessed metagenomic sequencing).
1D.iii.12 Intestinal Microbiome (Viruses) - Bray-Curtis dissimilarity | 12 months
  Measurement of beta diversity (assessed metagenomic sequencing).
1D.iv.0 Intestinal Microbiome (Viruses) - relative abundances of viruses. | Baseline
  ANCOM analysis (assessed metagenomic sequencing).
1D.iv.6 Intestinal Microbiome (Viruses) - relative abundances of viruses. | Change from baseline at 6 months
  ANCOM analysis (assessed metagenomic sequencing).
1D.iv.12 Intestinal Microbiome (Viruses) - relative abundances of viruses. | Change from baseline at 12 months
  ANCOM analysis (assessed metagenomic sequencing).
2A.i.0 Respiratory Microbiome (Bacteria) - Richness | Baseline
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.i.6 Respiratory Microbiome (Bacteria) - Richness | Change from baseline at 6 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.i.12 Respiratory Microbiome (Bacteria) - Richness | Change from baseline at 12 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.ii.0 Respiratory Microbiome (Bacteria) - Shannon index | Baseline
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.ii.6 Respiratory Microbiome (Bacteria) - Shannon index | Change from baseline at 6 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.ii.12 Respiratory Microbiome (Bacteria) - Shannon index | Change from baseline at 12 months
  Measurement of alpha diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.iii.0 Respiratory Microbiome (Bacteria) - UNIFRAC distances | Baseline
  Measurement of beta diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.iii.6 Respiratory Microbiome (Bacteria) - UNIFRAC distances | Change from baseline at 6 months
  Measurement of beta diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.iii.12 Respiratory Microbiome (Bacteria) - UNIFRAC distances | Change from baseline at 12 months
  Measurement of beta diversity (assessed using 16S rRNA or metagenomic gene sequencing).
2A.iv.0 Respiratory Microbiome (Bacteria) - relative abundances of bacteria | Baseline
  ANCOM analysis (assessed using 16S rRNA or metagenomic gene sequencing).
2A.iv.6 Respiratory Microbiome (Bacteria) - relative abundances of bacteria | Change from baseline at 6 months
  ANCOM analysis (assessed using 16S rRNA or metagenomic gene sequencing).
2A.iv.12 Respiratory Microbiome (Bacteria) - relative abundances of bacteria | Change from baseline at 12 months
  ANCOM analysis (assessed using 16S rRNA or metagenomic gene sequencing).
2B.i.0 Respiratory Microbiome (Proteome) - normalised abundances of proteins | Baseline
  (assessed using LC-MS).
2B.i.6 Respiratory Microbiome (Proteome) - normalised abundances of proteins | Change from baseline at 6 months
  (assessed using LC-MS).
2B.i.12 Respiratory Microbiome (Proteome) - normalised abundances of proteins | Change from baseline at 12 months
  (assessed using LC-MS).
2C.i.0 Respiratory Microbiome (Metabolome) - normalised abundances of metabolites | Baseline
  (assessed using LC-MS).
2C.i.6 Respiratory Microbiome (Metabolome) - normalised abundances of metabolites | Change from baseline at 6 months
  (assessed using LC-MS).
2C.i.12 Respiratory Microbiome (Metabolome) - normalised abundances of metabolites | Change from baseline at 12 months
  (assessed using LC-MS).
2D.i.0 Respiratory Microbiome (Viruses) - Richness | Baseline
  Measurement of alpha diversity (assessed metagenomic sequencing).
2D.i.6 Respiratory Microbiome (Viruses) - Richness | Change from baseline at 6 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
2D.i.12 Respiratory Microbiome (Viruses) - Richness | Change from baseline at 12 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
2D.ii.0 Respiratory Microbiome (Viruses) - Shannon index | Baseline
  Measurement of alpha diversity (assessed metagenomic sequencing).
2D.ii.6 Respiratory Microbiome (Viruses) - Shannon index | Change from baseline at 6 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
2D.ii.12 Respiratory Microbiome (Viruses) - Shannon index | Change from baseline at 12 months
  Measurement of alpha diversity (assessed metagenomic sequencing).
2D.iii.0 Respiratory Microbiome (Viruses) - Bray-Curtis dissimilarity | Baseline
  Measurement of beta diversity (assessed metagenomic sequencing).
2D.iii.6 Respiratory Microbiome (Viruses) - Bray-Curtis dissimilarity | 6 months
  Measurement of beta diversity (assessed metagenomic sequencing).
2D.iii.12 Respiratory Microbiome (Viruses) - Bray-Curtis dissimilarity | 12 months
  Measurement of beta diversity (assessed metagenomic sequencing).
2D.iv.0 Respiratory Microbiome (Viruses) - relative abundances of viruses | Baseline
  ANCOM analysis (assessed metagenomic sequencing).
2D.iv.6 Respiratory Microbiome (Viruses) - relative abundances of viruses | Change from baseline at 6 months
  ANCOM analysis (assessed metagenomic sequencing).
2D.iv.12 Respiratory Microbiome (Viruses) - relative abundances of viruses | Change from baseline at 12 months
  ANCOM analysis (assessed metagenomic sequencing).
3A.i.0 Diet - total energy intake | Baseline
  Kilojoules (assessed using a 24-hour recall or ACAES).
3A.i.6 Diet - total energy intake | Change from baseline at 6 months
  Kilojoules (assessed using a 24-hour recall or ACAES).
3A.i.12 Diet - total energy intake | Change from baseline at 12 months
  Kilojoules (assessed using a 24-hour recall or ACAES).
3B.i.0 Diet - percentage energy from core foods | Baseline
  (assessed using a 24-hour recall or ACAES).
3B.i.6 Diet - percentage energy from core foods | Change from baseline at 6 months
  (assessed using a 24-hour recall or ACAES).
3B.i.12 Diet - percentage energy from core foods | Change from baseline at 12 months
  (assessed using a 24-hour recall or ACAES).
3C.i.0 Diet - total macronutrients intake | Baseline
  Grams (assessed using a 24-hour recall or ACAES).
3C.i.6 Diet - total macronutrients intake | Change from baseline at 6 months
  Grams (assessed using a 24-hour recall or ACAES).
3C.i.12 Diet - total macronutrients intake | Change from baseline at 12 months
  Grams (assessed using a 24-hour recall or ACAES).
3C.ii.0 Diet - macronutrients proportion of total energy intake | Baseline
  Percentage (assessed using a 24-hour recall or ACAES).
3C.ii.6 Diet - macronutrients proportion of total energy intake | Change from baseline at 6 months
  Percentage (assessed using a 24-hour recall or ACAES).
3C.ii.12 Diet - macronutrients proportion of total energy intake | Change from baseline at 12 months
  Percentage (assessed using a 24-hour recall or ACAES).
3D.i.0 Diet - total micronutrients intake | Baseline
  Milligrams (assessed using a 24-hour recall or ACAES).
3D.i.6 Diet - total micronutrients intake | Change from baseline at 6 months
  Milligrams (assessed using a 24-hour recall or ACAES).
3D.i.12 Diet - total micronutrients intake | Change from baseline at 12 months
  Milligrams (assessed using a 24-hour recall or ACAES).
3D.ii.0 Diet - micronutrients proportion of total energy intake | Baseline
  Percentage (assessed using a 24-hour recall or ACAES).
3D.ii.6 Diet - micronutrients proportion of total energy intake | Change from baseline at 6 months
  Percentage (assessed using a 24-hour recall or ACAES).
3D.ii.12 Diet - micronutrients proportion of total energy intake | Change from baseline at 12 months
  Percentage (assessed using a 24-hour recall or ACAES).
3E.i.0 Diet - diet quality score | Baseline
  Australia recommended food score. Maximum possible score of 73, higher is better (assessed using the ACAES only).
3E.i.6 Diet - diet quality score | Change from baseline at 6 months
  Australia recommended food score. Maximum possible score of 73, higher is better (assessed using the ACAES only).
3E.i.12 Diet - diet quality score | Change from baseline at 12 months
  Australia recommended food score. Maximum possible score of 73, higher is better (assessed using the ACAES only).

SECONDARY OUTCOMES:
4A.i.0 Faecal biomarkers - calprotectin | Baseline
  mg/kg (assessed using an ELISA).
4A.i.6 Faecal biomarkers - calprotectin | Change from baseline at 6 months
  mg/kg (assessed using an ELISA).
4A.i.12 Faecal biomarkers - calprotectin | Change from baseline at 12 months
  mg/kg (assessed using an ELISA).
4A.ii.0 Faecal biomarkers - M2 pyruvate kinase | Baseline
  U/mL (assessed using an ELISA).
4A.ii.6 Faecal biomarkers - M2 pyruvate kinase | Change from baseline at 6 months
  U/mL (assessed using an ELISA).
4A.ii.12 Faecal biomarkers - M2 pyruvate kinase | Change from baseline at 12 months
  U/mL (assessed using an ELISA).
4A.iii.0 Faecal biomarkers - C-reactive protein | Baseline
  mg/L (assessed using an ELISA).
4A.iii.6 Faecal biomarkers - C-reactive protein | Change from baseline at 6 months
  mg/L (assessed using an ELISA).
4A.iii.12 Faecal biomarkers - C-reactive protein | Change from baseline at 12 months
  mg/L (assessed using an ELISA).
4A.iv.0 Faecal biomarkers - Interleukins | Baseline
  IU (assessed using an ELISA).
4A.iv.6 Faecal biomarkers - Interleukins | Change from baseline at 6 months
  IU (assessed using an ELISA).
4A.iv.12 Faecal biomarkers - Interleukins | Change from baseline at 12 months
  IU (assessed using an ELISA).
4B.i.0 Respiratory biomarkers - calprotectin | Baseline
  mg/kg (assessed using an ELISA).
4B.i.6 Respiratory biomarkers - calprotectin | Change from baseline at 6 months
  mg/kg (assessed using an ELISA).
4B.i.12 Respiratory biomarkers - calprotectin | Change from baseline at 12 months
  mg/kg (assessed using an ELISA).
4B.ii.0 Respiratory biomarkers - C-reactive protein | Baseline
  mg/L (assessed using an ELISA).
4B.ii.6 Respiratory biomarkers - C-reactive protein | Change from baseline at 6 months
  mg/L (assessed using an ELISA).
4B.ii.12 Respiratory biomarkers - C-reactive protein | Change from baseline at 12 months
  mg/L (assessed using an ELISA).
4B.iii.0 Respiratory biomarkers - Interleukins | Baseline
  IU (assessed using an ELISA).
4B.iii.6 Respiratory biomarkers - Interleukins | Change from baseline at 6 months
  IU (assessed using an ELISA).
4B.iii.12 Respiratory biomarkers - Interleukins | Change from baseline at 12 months
  IU (assessed using an ELISA).
5A.i.0 Symptomatology & HRQOL - PedsQL Infant Scales (ages 1-12 and 13-24 months) | Baseline
  Parent report for infants (ages 1-12 months) or (ages 13-24 months). Score out of 100, higher scores indicate better HRQOL.
5A.i.6 Symptomatology & HRQOL - PedsQL Infant Scales (ages 1-12 and 13-24 months) | Change from baseline at 6 months
  Parent report for infants (ages 1-12 months) or (ages 13-24 months). Score out of 100, higher scores indicate better HRQOL.
5A.i.12 Symptomatology & HRQOL - PedsQL Infant Scales (ages 1-12 and 13-24 months) | Change from baseline at 12 months
  Parent report for infants (ages 1-12 months) or (ages 13-24 months). Score out of 100, higher scores indicate better HRQOL.
5A.ii.0 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 2-4 years) | Baseline
  Parent report for toddlers (ages 2-4 years). Score out of 100, higher scores indicate better HRQOL.
5A.ii.6 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 2-4 years) | Change from baseline at 6 months
  Parent report for toddlers (ages 2-4 years). Score out of 100, higher scores indicate better HRQOL.
5A.ii.12 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 2-4 years) | Change from baseline at 12 months
  Parent report for toddlers (ages 2-4 years). Score out of 100, higher scores indicate better HRQOL.
5A.iii.0 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 5-7 years) | Baseline
  Parent report for young children (ages 5-7 years) or young child report (ages 5-7 years). Score out of 100, higher scores indicate better HRQOL.
5A.iii.6 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 5-7 years) | Change from baseline at 6 months
  Parent report for young children (ages 5-7 years) or young child report (ages 5-7 years). Score out of 100, higher scores indicate better HRQOL.
5A.iii.12 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 5-7 years) | Change from baseline at 12 months
  Parent report for young children (ages 5-7 years) or young child report (ages 5-7 years). Score out of 100, higher scores indicate better HRQOL.
5A.iv.0 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 8-12 years) | Baseline
  Parent report for children (ages 8-12 years) or child report (ages 8-12 years). Score out of 100, higher scores indicate better HRQOL.
5A.iv.6 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 8-12 years) | Change from baseline at 6 months
  Parent report for children (ages 8-12 years) or child report (ages 8-12 years). Score out of 100, higher scores indicate better HRQOL.
5A.iv.12 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 8-12 years) | Change from baseline at 12 months
  Parent report for children (ages 8-12 years) or child report (ages 8-12 years). Score out of 100, higher scores indicate better HRQOL.
5A.v.0 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 13-18 years) | Baseline
  Parent report for teens (ages 13-18 years) or teen report (ages 13-18 years). Score out of 100, higher scores indicate better HRQOL.
5A.v.6 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 13-18 years) | Change from baseline at 6 months
  Parent report for teens (ages 13-18 years) or teen report (ages 13-18 years). Score out of 100, higher scores indicate better HRQOL.
5A.v.12 Symptomatology & HRQOL - PedsQL Gastrointestinal Symptoms Module (ages 13-18 years) | Change from baseline at 12 months
  Parent report for teens (ages 13-18 years) or teen report (ages 13-18 years). Score out of 100, higher scores indicate better HRQOL.
5B.i.0 Symptomatology & HRQOL - Rome IV Parent-Report Form for Infants and Toddlers (ages 0-3) | Baseline
  29 items for ages 0-12 months. 18 items for ages 1-3 years. Defined diagnostic criteria for functional gastrointestinal disorders in neonates and toddlers: Infant regurgitation, Infant rumination syndrome, Cyclic vomiting syndrome, Infant colic, Functional diarrhoea, Infant dyschezia, Functional constipation.
5B.i.6 Symptomatology & HRQOL - Rome IV Parent-Report Form for Infants and Toddlers (ages 0-3) | 6 months
  29 items for ages 0-12 months. 18 items for ages 1-3 years. Defined diagnostic criteria for functional gastrointestinal disorders in neonates and toddlers: Infant regurgitation, Infant rumination syndrome, Cyclic vomiting syndrome, Infant colic, Functional diarrhoea, Infant dyschezia, Functional constipation.
5B.i.12 Symptomatology & HRQOL - Rome IV Parent-Report Form for Infants and Toddlers (ages 0-3) | 12 months
  29 items for ages 0-12 months. 18 items for ages 1-3 years. Defined diagnostic criteria for functional gastrointestinal disorders in neonates and toddlers: Infant regurgitation, Infant rumination syndrome, Cyclic vomiting syndrome, Infant colic, Functional diarrhoea, Infant dyschezia, Functional constipation.
5B.ii.0 Symptomatology & HRQOL - Rome IV Parent-Report Form for Children and Adolescents (4 years of age and older) | Baseline
  42 items. Defined diagnostic criteria for functional gastrointestinal disorders in children and adolescents: Cyclic vomiting syndrome, Functional nausea and functional vomiting, Rumination syndrome, Aerophagia, Functional dyspepsia, Irritable bowel syndrome, Abdominal migraine, Functional abdominal pain - not otherwise specified, Functional Constipation, Nonretentive fecal incontinence.
5B.ii.6 Symptomatology & HRQOL - Rome IV Parent-Report Form for Children and Adolescents (4 years of age and older) | 6 months
  42 items. Defined diagnostic criteria for functional gastrointestinal disorders in children and adolescents: Cyclic vomiting syndrome, Functional nausea and functional vomiting, Rumination syndrome, Aerophagia, Functional dyspepsia, Irritable bowel syndrome, Abdominal migraine, Functional abdominal pain - not otherwise specified, Functional Constipation, Nonretentive fecal incontinence.
5B.ii.12 Symptomatology & HRQOL - Rome IV Parent-Report Form for Children and Adolescents (4 years of age and older) | 12 months
  42 items. Defined diagnostic criteria for functional gastrointestinal disorders in children and adolescents: Cyclic vomiting syndrome, Functional nausea and functional vomiting, Rumination syndrome, Aerophagia, Functional dyspepsia, Irritable bowel syndrome, Abdominal migraine, Functional abdominal pain - not otherwise specified, Functional Constipation, Nonretentive fecal incontinence.
5B.iii.0 Symptomatology & HRQOL - Rome IV Self-Report Form for Children and Adolescents (10 years of age and older) | Baseline
  42 items. Defined diagnostic criteria for functional gastrointestinal disorders in children and adolescents: Cyclic vomiting syndrome, Functional nausea and functional vomiting, Rumination syndrome, Aerophagia, Functional dyspepsia, Irritable bowel syndrome, Abdominal migraine, Functional abdominal pain - not otherwise specified, Functional Constipation, Nonretentive fecal incontinence.
5B.iii.6 Symptomatology & HRQOL - Rome IV Self-Report Form for Children and Adolescents (10 years of age and older) | 6 months
  42 items. Defined diagnostic criteria for functional gastrointestinal disorders in children and adolescents: Cyclic vomiting syndrome, Functional nausea and functional vomiting, Rumination syndrome, Aerophagia, Functional dyspepsia, Irritable bowel syndrome, Abdominal migraine, Functional abdominal pain - not otherwise specified, Functional Constipation, Nonretentive fecal incontinence.
5B.iii.12 Symptomatology & HRQOL - Rome IV Self-Report Form for Children and Adolescents (10 years of age and older) | 12 months
  42 items. Defined diagnostic criteria for functional gastrointestinal disorders in children and adolescents: Cyclic vomiting syndrome, Functional nausea and functional vomiting, Rumination syndrome, Aerophagia, Functional dyspepsia, Irritable bowel syndrome, Abdominal migraine, Functional abdominal pain - not otherwise specified, Functional Constipation, Nonretentive fecal incontinence.
5C.i.0 Symptomatology & HRQOL - Spence Children's Anxiety Scale; Preschool Anxiety Scale (Parent report for ages 0 to 4) | Baseline
  34 items. Maximum possible scores of 112. A score 1 SD above mean for a subscale or total score warrants further clinical investigation. A score of 0.5 SD above the mean on total score is indicative of an elevated, but not clinical level of anxiety.
5C.i.6 Symptomatology & HRQOL - Spence Children's Anxiety Scale; Preschool Anxiety Scale (Parent report for ages 0 to 4) | Change from baseline at 6 months
  34 items. Maximum possible scores of 112. A score 1 SD above mean for a subscale or total score warrants further clinical investigation. A score of 0.5 SD above the mean on total score is indicative of an elevated, but not clinical level of anxiety.
5C.i.12 Symptomatology & HRQOL - Spence Children's Anxiety Scale; Preschool Anxiety Scale (Parent report for ages 0 to 4) | Change from baseline at 12 months
  34 items. Maximum possible scores of 112. A score 1 SD above mean for a subscale or total score warrants further clinical investigation. A score of 0.5 SD above the mean on total score is indicative of an elevated, but not clinical level of anxiety.
5C.ii.0 Symptomatology & HRQOL - Spence Children's Anxiety Scale (Parent report for 5 years and older) | Baseline
  38 scored items. Maximum possible scores of 114. A score 1 SD above mean (T-score of ≥ 60) for a subscale or total score is indicative of subclinical or elevated levels of anxiety warranting further clinical investigation.
5C.ii.6 Symptomatology & HRQOL - Spence Children's Anxiety Scale (Parent report for 5 years and older) | Change from baseline at 6 months
  38 scored items. Maximum possible scores of 114. A score 1 SD above mean (T-score of ≥ 60) for a subscale or total score is indicative of subclinical or elevated levels of anxiety warranting further clinical investigation.
5C.ii.12 Symptomatology & HRQOL - Spence Children's Anxiety Scale (Parent report for 5 years and older) | Change from baseline at 12 months
  38 scored items. Maximum possible scores of 114. A score 1 SD above mean (T-score of ≥ 60) for a subscale or total score is indicative of subclinical or elevated levels of anxiety warranting further clinical investigation.
5C.iii.0 Symptomatology & HRQOL - Spence Children's Anxiety Scale (8 years and older) | Baseline
  38 scored items. Maximum possible scores of 114. A score 1 SD above mean (T-score of ≥ 60) for a subscale or total score is indicative of subclinical or elevated levels of anxiety warranting further clinical investigation.
5C.iii.6 Symptomatology & HRQOL - Spence Children's Anxiety Scale (8 years and older) | Change from baseline at 6 months
  38 scored items. Maximum possible scores of 114. A score 1 SD above mean (T-score of ≥ 60) for a subscale or total score is indicative of subclinical or elevated levels of anxiety warranting further clinical investigation.
5C.iii.12 Symptomatology & HRQOL - Spence Children's Anxiety Scale (8 years and older) | Change from baseline at 12 months
  38 scored items. Maximum possible scores of 114. A score 1 SD above mean (T-score of ≥ 60) for a subscale or total score is indicative of subclinical or elevated levels of anxiety warranting further clinical investigation.
5D.i.0 Symptomatology & HRQOL - Mood and Feelings Questionnaire (Short Version) (Parent Report on Child, ages 6-18 years). | Baseline
  13 items. Maximum possible scores of 26. Higher scores suggest more severe depressive symptoms. A score of ≥ 12 may indicate the presence of depression in the respondent.
5D.i.6 Symptomatology & HRQOL - Mood and Feelings Questionnaire (Short Version) (Parent Report on Child, ages 6-18 years). | Change from baseline at 6 months
  13 items. Maximum possible scores of 26. Higher scores suggest more severe depressive symptoms. A score of ≥ 12 may indicate the presence of depression in the respondent.
5D.i.12 Symptomatology & HRQOL - Mood and Feelings Questionnaire (Short Version) (Parent Report on Child, ages 6-18 years). | Change from baseline at 12 months
  13 items. Maximum possible scores of 26. Higher scores suggest more severe depressive symptoms. A score of ≥ 12 may indicate the presence of depression in the respondent.
5D.ii.0 Symptomatology & HRQOL - Mood and Feelings Questionnaire (Short Version) (Child Self Report, ages 6-18 years). | Baseline
  13 items. Maximum possible scores of 26. Higher scores suggest more severe depressive symptoms. A score of ≥ 12 may indicate the presence of depression in the respondent.
5D.ii.6 Symptomatology & HRQOL - Mood and Feelings Questionnaire (Short Version) (Child Self Report, ages 6-18 years). | Change from baseline at 6 months
  13 items. Maximum possible scores of 26. Higher scores suggest more severe depressive symptoms. A score of ≥ 12 may indicate the presence of depression in the respondent.
5D.ii.12 Symptomatology & HRQOL - Mood and Feelings Questionnaire (Short Version) (Child Self Report, ages 6-18 years). | Change from baseline at 12 months
  13 items. Maximum possible scores of 26. Higher scores suggest more severe depressive symptoms. A score of ≥ 12 may indicate the presence of depression in the respondent.
6A.i.0 Phenotypic & Clinical Information - Weight (ages 0 to 20 years) | Baseline
  Z-score.
6A.i.6 Phenotypic & Clinical Information - Weight (ages 0 to 20 years) | Change from baseline at 6 months
  Z-score.
6A.i.12 Phenotypic & Clinical Information - Weight (ages 0 to 20 years) | Change from baseline at 12 months
  Z-score.
6A.ii.0 Phenotypic & Clinical Information - Length (ages 0 to 2 years) | Baseline
  Z-score.
6A.ii.6 Phenotypic & Clinical Information - Length (ages 0 to 2 years) | Change from baseline at 6 months
  Z-score.
6A.ii.12 Phenotypic & Clinical Information - Length (ages 0 to 2 years) | Change from baseline at 12 months
  Z-score.
6A.iii.0 Phenotypic & Clinical Information - Height (ages 2 to 20 years) | Baseline
  Z-score.
6A.iii.6 Phenotypic & Clinical Information - Height (ages 2 to 20 years) | Change from baseline at 6 months
  Z-score.
6A.iii.12 Phenotypic & Clinical Information - Height (ages 2 to 20 years) | Change from baseline at 12 months
  Z-score.
6A.iv.0 Phenotypic & Clinical Information - Weight-for-length (ages 0 to 2 years) | Baseline
  Z-score.
6A.iv.6 Phenotypic & Clinical Information - Weight-for-length (ages 0 to 2 years) | Change from baseline at 6 months
  Z-score.
6A.iv.12 Phenotypic & Clinical Information - Weight-for-length (ages 0 to 2 years) | Change from baseline at 12 months
  Z-score.
6A.v.0 Phenotypic & Clinical Information - Body mass index (ages 2 to 20 years) | Baseline
  Z-score.
6A.v.6 Phenotypic & Clinical Information - Body mass index (ages 2 to 20 years) | Change from baseline at 6 months
  Z-score.
6A.v.12 Phenotypic & Clinical Information - Body mass index (ages 2 to 20 years) | Change from baseline at 12 months
  Z-score.
6B.i.6 Phenotypic & Clinical Information - Number of hospitalisations | 6 months
  During period from baseline to 6 months.
6B.i.12 Phenotypic & Clinical Information - Number of hospitalisations | 12 months
  During period from baseline to 12 months.
6B.ii.6 Phenotypic & Clinical Information - Length of hospitalisations | 6 months
  Days hospitalised during period from baseline to 6 months.
6B.ii.12 Phenotypic & Clinical Information - Length of hospitalisations | 12 months
  Days hospitalised during period from baseline to 12 months.
6B.iii.6 Phenotypic & Clinical Information - Number of emergency department presentations | 6 months
  During period from baseline to 6 months.
6B.iii.12 Phenotypic & Clinical Information - Number of emergency department presentations | 12 months
  During period from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Coffey, Principal Investigator — University of New South Wales; Chee (Keith) Y Ooi, Principal Investigator — University of New South Wales
Locations (1):
- Sydney Children's Hospital, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
De-identified data and biological samples may be utilised by study investigators ONLY for the sole purpose of a research project.

REFERENCES:
- [Derived] McKay I, van Dorst J, Katz T, Doumit M, Prentice B, Owens L, Belessis Y, Chuang S, Jaffe A, Thomas T, Coffey M, Ooi CY. Diet and the gut-lung axis in cystic fibrosis - direct & indirect links. Gut Microbes. 2023 Jan-Dec;15(1):2156254. doi: 10.1080/19490976.2022.2156254. PMID 36573804
- [Derived] Traini I, Chan SY, Menzies J, Hughes J, Coffey MJ, Katz T, McKay IR, Ooi CY, Leach ST, Krishnan U. Evaluating the Dietary Intake of Children With Esophageal Atresia: A Prospective, Controlled, Observational Study. J Pediatr Gastroenterol Nutr. 2022 Aug 1;75(2):221-226. doi: 10.1097/MPG.0000000000003498. Epub 2022 Jun 1. PMID 35653431
- [Derived] Coffey MJ, McKay IR, Doumit M, Chuang S, Adams S, Stelzer-Braid S, Waters SA, Kasparian NA, Thomas T, Jaffe A, Katz T, Ooi CY. Evaluating the Alimentary and Respiratory Tracts in Health and disease (EARTH) research programme: a protocol for prospective, longitudinal, controlled, observational studies in children with chronic disease at an Australian tertiary paediatric hospital. BMJ Open. 2020 Apr 14;10(4):e033916. doi: 10.1136/bmjopen-2019-033916. PMID 32295774